CLINICAL TRIAL: NCT05545670
Title: Allopurinol Impact on Cirrhosis Related Complications
Brief Title: Allopurinol to Prevent Cirrhosis Related Morbidities
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Khadija Ahmed Mhrose Glal, assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: allopurinol in cirrhosis
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Group1: (Placebo, n=50) who will receive oral placebo tablet once daily FOR 6 MONTHS
  Interventions: Drug: Placebo
- allopurinol (Active Comparator): Group 2:(Allopurinol n=50) who will receive oral allopurinol 300 mg daily for 6 months
  Interventions: Drug: Allopurinol 300 MG

INTERVENTIONS:
Drug: Placebo — not containing drugs
  Arms: placebo
Drug: Allopurinol 300 MG — a competitive xanthine oxidase inhibitor, reduces oxidative stress and attenuates bacterial translocation
  Arms: allopurinol

SUMMARY:
The study aims to compare the potential benefit of allopurinol in reducing the risk of developing cirrhosis-related complications, delaying the onset of hepatocellular carcinoma, and improving survival. Furthermore, the study aims to evaluate their impact on parents' related quality of life

DETAILED DESCRIPTION:
Cirrhosis is the late stage of liver damage and possess two phases: a compensated phase with favorable prognosis and a decompensated phase with high mortality rate.The shift from compensated to decompensated cirrhosis is characterized by the onset of complications, including ascites, hepatic encephalopathy (HE), variceal bleeding, and spontaneous bacterial peritonitis (SBP) which are associated with substantial morbidity and negative Impact on quality of life (QOL).

The gut microbiota plays an important role in cirrhosis and development of cirrhosis-related complications.

Indeed, translocation of endotoxins is increased in patients with cirrhosis and patients with more severe cirrhosis (i.e. Patients with decompensated cirrhosis, hospitalized patients) had significantly greater serum endotoxin concentrations that mediate complications of cirrhosis.

Intestinal permeability plays a role in the development of bacterial translocation and may be involved in the development of complications of cirrhosis. This 'leaky gut' phenomenon increases with the degree of liver failure and is particularly prominent in patients with cirrhosis who have experienced severe septic complications and has been implicated in the hepatic production of endotoxin-associated proinflammatory cytokines.

Intestinal mucosa alterations at the subcellular level have been reported in experimental cirrhosis, in relation to an increased oxidative stress due to overactivity in the enzyme xanthine oxidase.

Allopurinol, a competitive xanthine oxidase inhibitor, reduces oxidative stress and attenuates bacterial translocation in portal hypertensive animals, suggesting that the damaging effects of oxygen-derived free radicals and peroxidation on mucosal cells may be counteracted by a free radical scavenger.

In 2007, a pilot study demonstrated that allopurinol in patients with cirrhosis is associated with a significant reduction in oxidative stress but no effect on intestinal permeability and inflammatory markers. The study duration was only 10 days and therefore another study with a long period of time is essential.

ELIGIBILITY:
Inclusion Criteria:

* ge 18 to 75 years old Both sex Adults with cirrhosis in a stable conditions

Exclusion Criteria:

* Active SBP Renal insufficiency (serum creatinine > 2.0 mg/dl) Active GIT hemorrhage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
morbidities | 6 moths
  occurrence or exacerbation of complication

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Glal KAM, El-Haggar SM, Abdel-Salam SM, Mostafa TM. Allopurinol Prevents Cirrhosis-Related Complications: A Quadruple Blind Placebo-Controlled Trial. Am J Med. 2024 Jan;137(1):55-64. doi: 10.1016/j.amjmed.2023.09.016. Epub 2023 Oct 12. PMID 37832758